CLINICAL TRIAL: NCT00495196
Title: Cardiovascular Response to Peripheral Chemoreceptor Stimulation in Congestive Heart Failure With Cheyne- Stokes Respiration
Brief Title: Cardiovascular Responses in Congestive Heart Failure With Cheyne- Stokes Respiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Rachel Coxon, ResMed
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: X07-0079
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Heart Failure, Congestive; Cheyne-Stokes Respiration
MeSH Terms: conditions — Heart Failure; Cheyne-Stokes Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Experimental lung function test
- 2 (Active Comparator)
  Interventions: Procedure: Experimental lung function test

INTERVENTIONS:
Procedure: Experimental lung function test — Administration of several CO2 gas mixtures

SUMMARY:
The purpose of the trial is to investigate the cardiovascular response to peripheral chemoreceptor stimulation in Congestive Heart Failure with Cheyne- Stokes Respiration

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe heart failure (NYHA Class II or above) on optimal medical therapy
* LVEF less than or equal to 45%
* Stable condition as defined as no hospital admission or changes to medical therapy within two weeks prior to enrolment

Exclusion Criteria:

* Patients taking known respiratory stimulants or depressants
* Clinically significant asthma requiring therapy
* Significant parenchymal lung disease
* Primary pulmonary hypertension
* Myocardial infarction within three months prior to enrolment
* Patients with cardiac resynchronisation devices and permanent pacemakers
* Anaemic (haemoglobin < 12g/dL)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular parameters such as continuous blood pressure and heart rate. | During administration of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Coxon, BE/MBiomedE, Study Director — ResMed/The University of New South Wales; Klaus Schindhelm, PhD, Study Director — ResMed/The University of New South Wales; Jodie Lattimore, PhD, Study Director — Royal Prince Alfred Hospital, Sydney, Australia; Ian Wilcox, PhD, Principal Investigator — Royal Prince Alfred Hospital/The University of Sydney
Locations (1):
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia